CLINICAL TRIAL: NCT01261702
Title: Intravenous Magnesium Infusion for Pain Relief After Thoracotomy. A Randomized Controlled Trial.
Brief Title: Magnesium Infusion for Pain Relief After Thoracotomy. A Randomized Controlled Trial.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: not include patient anymore
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 008/2552
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Magnesium Sulphate; Post Pulmonary Resection; Pain
Keywords: Magnesium sulphate; Post Pulmonary Resection; Pain
MeSH Terms: conditions — Pain | interventions — Magnesium Sulfate; Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline IV
  Interventions: Drug: Placebo
- Magnesium sulphate (Experimental): Magnesium sulphate 50 mg/kg of magnesium sulphate infusion in 10 minutes before induction and then 15 mg/kg/hr until the end of the surgery.
  Interventions: Drug: magnesium sulphate

INTERVENTIONS:
Drug: Placebo — Normal saline IV
  Other Names: NSS
  Arms: Placebo
Drug: magnesium sulphate — The magnesium group (Group M, n=16) received 50 mg/kg of magnesium sulphate infusion in 10 minutes before induction and then 15 mg/kg/hr until the end of the surgery.
  Other Names: magnesium
  Arms: Magnesium sulphate

SUMMARY:
All patients were premedicated with oral midazolam 5-15 mg. one hour before surgery. General anesthesia with double lumen endobronchial tube was given. Patient was induced by propofol and fentanyl. Cisatracurium was given to facilitate intubation. Patient was ventilated with 50% oxygen in air. Anesthesia was maintained with propofol and fentanyl in order to keep blood pressure and heart rate within 20% of the baseline. Cisatracurium was given every 30 minutes in order to control ventilation. At the end of surgery, neuromuscular blockade was reversed.In PACU, the I.V. PCA machine was connected to the patient. The setting of PCA was basal infusion of morphine 1 mg/hr bolus of morphine 1 mg with lockout interval 5 minutes and 4-hour limit 30 mg.The patient's mean arterial blood pressure, heart rate were recorded before induction, before intubation, at 15, 15, 30, 60, 90 and 120 minutes after intubation, and at 4, 8,16 and 24 h after surgery. The total amounts of fentanyl, propofol and magnesium sulphate were recorded. The time between the cessation of magnesium sulphate and extubation was recorded. The amounts of morphine usage at 4, 8, 16 and 24 hours after surgery were recorded. Pain score was evaluated at rest and deep breath and sedation score at 1, 2, 3, 4, 8, 16 and 24 hours after surgery using numeric rating scale (NRS). Sedation score was graded as 0 = fully awake, 1 = somnolence, responds to call, 2 = somnolence, responds to tactile stimulation, 3 = asleep, responds to painful stimulation. The times that the patient first sipping, taking food, sitting at the edge of bed and walk with help were also recorded. The side effects such as nausea, vomiting, pruritus and respiratory depression were recorded. Cost effective analysis was also evaluated.

DETAILED DESCRIPTION:
All patients were premedicated with oral midazolam 5-15 mg. one hour before surgery. In the operating room, each patient was monitored with noninvasive blood pressure, ECG and pulse oximetry. After the patient was anesthetized, direct blood pressure, end-tidal carbon dioxide tension (ETCO2) and esophageal temperature were monitored. Choice of anesthesia was general anesthesia with double lumen endobronchial tube (Bronchocath). Patient was induced by propofol 1.5-2.5 mg/kg and fentanyl 2 μg/kg. After the patient was unconscious, cisatracurium 0.2 mg/kg was given to facilitate intubation. Patient was ventilated with 50% oxygen in air. Anesthesia was maintained with propofol 6 -12 mg/kg/hr and 1 μg/kg of fentanyl was given intermittently every 1-1.5 hour in order to keep blood pressure and heart rate within 20% of the baseline. Cisatracurium (0.03 mg/kg) was given every 30 minutes in order to control ventilation. The patient was ventilated with volume controlled ventilator. Throughout the surgery, the ETCO2 was kept between 30-35 mmHg. During two lung ventilation, the airway pressure was kept within 20 cmH2O and respiratory rate 10-12 beats/minute. One lung ventilation was achieved with airway pressure less than 30 cmH2O and respiratory rate 12-20 beats/minute. During the surgery, the lower part of the patient was warmed with forced air warmer (Bier Hugger) At the end of surgery, neuromuscular blockade was reversed by prostigmine 2.5 mg and atropine 1.2 mg.

In the post anesthesia care unit, the I.V. PCA machine was connected to the patient. The setting of PCA was basal infusion of morphine 1 mg/hr bolus of morphine 1 mg with lockout interval 5 minutes and 4-hour limit 30 mg. The patient's mean arterial blood pressure, heart rate were recorded before induction, before intubation, at 15, 15, 30, 60, 90 and 120 minutes after intubation, and at 4, 8 , 16 and 24 hour after surgery. The total amounts of fentanyl, propofol and magnesium sulphate were recorded. The time between the cessation of magnesium sulphate and extubation was recorded. The amounts of morphine usage at 4, 8, 16 and 24 hours after surgery were recorded. Pain score was evaluated at rest and deep breath and sedation score at 1, 2, 3, 4, 8, 16 and 24 hours after surgery using numeric rating scale (NRS). Sedation score was graded as 0 = fully awake, 1 = somnolence, responds to call, 2 = somnolence, responds to tactile stimulation, 3 = asleep, responds to painful stimulation. The times that the patient first sipping, taking food, sitting at the edge of bed and walk with help were also recorded. The side effects such as nausea, vomiting, pruritus and respiratory depression were recorded. Cost effective analysis was also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* Age 18-65 year
* ASA physical status 1-3
* Can use patient-controlled analgesia (PCA)

Exclusion Criteria:

* History of allergy to magnesium sulphate
* History of COPD, asthma or liver disease
* Serum creatinine > 1.5 mg/dL
* History of CHF or atrioventricular conduction disturbance
* History of taking calcium channel blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Total 24 hour morphine requirement | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Charroonpong Choorat, Ubon Ratchathani, Thailand